CLINICAL TRIAL: NCT00695799
Title: Measurement Of Propofol Concentration In The Ambient Air Of The Operating Room And In The Blood Of Anesthesia Care Providers During Propofol -Based General Anesthesia
Brief Title: Propofol Concentration In The Ambient Air Of The Operating Room And In The Blood Of Anesthesia Care Providers
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Anesthesia, Ming Xiong, MD, Associate Professor, Rutgers, The State University of New Jersey
Other Study IDs: 0120080063
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Propofol Pollution
Keywords: Propofol; Anesthesia care provider; Pollution; Operating room; Environment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Standard blood draw
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Anesthesia Providers at UMDNJ

SUMMARY:
The pollution of the operating room environment by anesthetic agents had been questioned, studied and documented in the past. These investigations demonstrated the existence of teratogenic effects in animals and the possibility of a decrease in mental performance, reduced fertility, fetal loss, spontaneous abortion and addictive potential in humans with chronic exposure to trace amounts of anesthetic agents. These findings led to the establishment of exposure limits and industry standards by consumer protection agencies, such as National Institute for Occupational Safety and Health (NIOSH). However, these standards applied to inhalation anesthetic agents that were excreted from the lungs of patients during expiration. These concerns about operating room pollution weaned away with the introduction of intravenous anesthetic agents, such as propofol, because it was believed propofol was excreted by systems other than the lungs. Recent research points to the contrary and demonstrates the excretion of propofol vapor in the expired gases of patients. Furthermore, animal experiments in our laboratory establish the existence of a biological mechanism responsible for addiction in animals exposed to trace amounts of propofol. We propose to study the exposure levels of anesthesia care providers in the operating room, during propofol use, under standardized conditions. Our findings will help to establish preventive measures for propofol addiction in anesthesia care providers.

DETAILED DESCRIPTION:
This clinical project will be carried out in the operating rooms of the University Hospital and the Doctors Office Center. The study will be done during routine surgery where a laryngeal mask airway will be used to maintain airway during general anesthesia in 20 adult patients with American Society of Anesthesiologists physical status I or II. Routine anesthetic care standards will be applied in intravenous line placement and monitoring of patients. General anesthesia will be induced with a bolus dose of propofol (2mg.kg-1) and maintained with an intravenous infusion of propofol (100-200 mcg.kg-1.min-1). Patients will be allowed to breathe spontaneously 40% oxygen in air. Adjuvant intravenous medications will be given for amnesia, analgesia and infection prophylaxis as per routine anesthetic practice. The ambient propofol concentration will be measured, using a proton transfer reaction mass spectrometer (PTR-MS), at a distance of 25cm from the patient's face. The measurement of ambient propofol concentration will begin before the administration of propofol to the patient and will continue till the patient leaves the operating room. The use of PTR-MS device will not interfere with the anesthetic management of patient. In an unforeseen circumstance, where the anesthesiologist determines the use of PTR-MS does interfere with the anesthetic care of the patient, the device will be immediately removed and the measurement of ambient propofol concentration will be suspended for the case. The set-up and usage of PTR-MS will be performed by a research team that does not take part in the clinical management of the patient. The PTR-MS is a device that depends on the proton transfer reaction to quantify, in parts per billion (ppb) by volume, volatile organic compounds in air at extremely low concentrations and in real time. The mean and peak ambient propofol concentration will be determined during each case and a time weighted average (TWA) will be calculated for an eight-hour period at the end of the study. In addition, after receiving written informed consent from anesthesia care providers, blood samples will be drawn from them and propofol concentrations will be measured by high-performance liquid chromatography (HPLC) within 24hr. The blood samples will constitute 3ml on two occasions, one early in the morning before anesthesia care starts and one after eight hours of anesthesia care. HPLC is a device that uses a spectrofluorometric detector to estimate trace amounts of propofol in blood in ng.ml-1. The blood estimation of propofol will also be conducted by a research team that does not take part in the clinical management of patients.

ELIGIBILITY:
Inclusion Criteria:

* If you are over the age of 18- and under 65, and mentally capable of giving consent.
* If you are an Anesthesiology staff member.
* If you are scheduled to administer propofol during general anesthesia and surgery

Exclusion Criteria:

* If you refuse to sign consent.
* If you are not administering propofol within 8 hours after your first blood draw.
* If you are pregnant.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Anesthesia care providers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Level of propofol in the air of the OR and blood of the anesthesia provider | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ming Xiong, PHD, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ, Newark, New Jersey, United States